CLINICAL TRIAL: NCT05523557
Title: Rehabilitation in Pulmonary Hypertension: Effects of an Urban-training Program.
Brief Title: Urban-training Intervention in Pulmonary Hypertension (UTHAP)
Acronym: UTHAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UrbanTrainHAP
Record Dates: First submitted 2022-08-16; First posted 2022-08-31 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urban Training Group (Experimental): The PA will consist of the following components: motivational interview, exercise following a dossier containing various maps of Urban Training walking trails (at least 30 minutes per day/5 days per week) and use of a Fitbit Inspire (FitBit, San Francisco) and motivational follow-up visit, in group, once per month during the follow-up period.
  Interventions: Behavioral: Urban Training
- Control Group (No Intervention): The intervention will consist of a general recommendation to perform regular physical activity .

INTERVENTIONS:
Behavioral: Urban Training — 1) one-to-one motivational interview for a maximum of 1h; 2) exercise following a dossier containing various maps of Urban Training walking trails, previously used in patients with COPD with a recommendation of doing a minimum of 1 circuit/day; or in case of living faraway from Urban Training walking trails, the instructions will be to walk at least 30 minutes per day ⩾5 days per week, at a pace reaching a dyspnoea Borg scale score of 4 -6; 3) a FitBit Inspire (FitBit, San Francisco, United States) to obtain direct feedback on the step count and intensity of PA; and 4) a motivational follow-up visit, in group, once per month during the follow-up period.
  Arms: Urban Training Group

SUMMARY:
Pulmonary rehabilitation is effective in the treatment of pulmonary hypertension (PH). However, the beneficial effects of such intervention have been seen to disappear over time in other chronic diseases. The objective of the project is to evaluate the efficacy of an urban exercise program after a rehabilitation program and to identify possible determinants of sustainability of the effect, both in patients and in a murine experimental model.

Methodology: 1) Study in humans: randomized study (urban training) in 80 patients with PH. The main variable is the improvement in physical activity measured by accelerometry at 12 months. Improvements in bioimpedance and aerobic capacity will be analysed as secondary variables, as well as possible determinants of vascular function that guarantee the sustainability of the effect (pulse wave velocity, endothelial function, metabolic profile and other plasma biomarkers), and all of them will be correlated with the evolution of the disease (admission due to clinical deterioration). 2) Studies in a murine experimental model: Mice with pulmonary hypertension induced by the administration of SU5416 (sugen) and exposure to hypoxia for 3 weeks will be studied after a three-week rehabilitation program. Half of them will exercise 1-2 days a week for 4 more weeks. At the end of the program, the right ventricular pressure will be measured and subsequently the animals will be sacrificed. Morphometric studies will be performed on lung, cardiac and muscular tissue. Vascular endothelial function and autophagy will be also measured. The differences in these variables between the different experimental groups will be analysed.

DETAILED DESCRIPTION:
Background Pulmonary arterial hypertension (PAH) and chronic thromboembolic pulmonary hypertension (CTEPH) are rare forms of PH (ORPHA 182090) that affect small pulmonary arteries and is characterized by gradual obliteration of arterial lumen. This results in a progressive increase in pulmonary vascular resistance that may eventually result in right ventricular failure and death. The disease carries a high mortality, especially if not treated properly, with a life expectancy of less than 3 years. In recent years there has been great progress in the study of the disease in the fields of genetics, pathophysiology and treatment of PAH. Thanks to that, the development of new drugs and treatment strategies has improved the prognosis of the disease and in most cases, has improved exercise tolerance. Importantly, complementary to the targeted pharmacological treatment of PAH, a series of actions are essentials to increase their effectiveness, including supportive treatments and general measures (preventing pregnancy, preventing infections, psychosocial support and exercise training).

Exercise-based pulmonary rehabilitation is widely recognized as a non-pharmacological strategy able to improve muscular function and exercise tolerance and reduce dyspnea in patients with PAH and CTEPH. At present, there are no recommendations on what to do to maintain the effects after a rehabilitation program or any tool that can be used in routine clinical practice to increase long-term effects or sustainability of the program. In summary, to guarantee the accomplishment of a certain degree of physical activity after a rehabilitation program, an urban training program emerges as a sustainable alternative.

The idea of an urban training program was born as an alternative of monitored in-hospital exercise training due to the difficulty to offer an intensive and maintained exercise medical care approach due to the increasing number of patients with chronic respiratory diseases, such as chronic obstructive pulmonary disease (COPD). These patients needed a sustained practice of physical activity, and the urban training program was supported by the fact that walking is a practice fully integrated into the daily lives of patients in Mediterranean countries. The current project proposes that the patients' usual walks can be adapted to the needs and abilities of their illness using public spaces and urban itineraries.

General study design Based on this background, the general purpose of the project is to implement an urban exercise program (sustainable) in patients with PAH and CTEPH with a double objective, first, to further extend the beneficial effects of the hospital rehabilitation program and second to investigate the physiological and molecular factors that determine the degree of this response. The project has a translational design in which the effects of exercise on vascular function will be studied both in patients with PAH or CTEPH and in an animal model of pulmonary hypertension. Two studies will be carried out, the first, in humans, where the phenotype of patients who show little efficacy and effectiveness of an urban training program will be characterized. The second, in a murine PH model (sugen + hypoxia in mice), a model developed and validated in a previous project of our group where the changes on the gene expression profile in the lung, heart and skeletal muscle will be evaluated after an exercise program. In the first study, clinical and functional response of patients diagnosed and monitored in our centre for PAH and CTEPH, who had completed a 3-month physical exercise program, will be evaluated, one year after the end of the program with an urban intervention training that will last a maximum of one year, compared with usual care. Similarly, vascular function, impedance measurement, as well as other functional and metabolic parameters will be analysed before and after one year in order to identify parameters that ensure the sustainability of the effects achieved after the rehabilitation program. In the second study, we will analyze in mice, after a treadmill program, the main molecular pathways activated or inhibited by physical exercise. In this study we will perform a differential analysis of gene expression in different tissues (lung, heart and muscle) and a in-silico analysis with the objective to identify new biomarkers of functional status (lung, heart and muscle function). Validated results in this animal model could be tested in a next step in blood samples from patients with PAH or CTEPH.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* New York Health Association (NYHA) II-III functional class;
* PAH or CTEPH diagnosed by right heart catheterization, evidencing: mean pulmonary arterial pressure (PAPm) ≥25 mmHg; pulmonary wedge pressure (PCWP) ≤15 mmHg; and pulmonary vascular resistance (PVR) ≥240 din/s/cm5 or 3 woods unit (WU);
* Patients with optimized PH targeted treatment, including intensified diuretic treatment and who have remained stable for at least 2 months before entering the study (no changes in medical treatment are expected throughout the 12-week study period);
* Patients who already finished a 3-months rehabilitation program;
* Be able to understand and be willing to sign the informed consent form.

Exclusion Criteria:

* Patients with other forms of PH (groups 2, 3 or 5);
* Pregnancy;
* Patients with signs of right heart decompensation;
* Inability to exercise on a cycle ergometer or walking;
* Acute infection or fever;
* Any change in the treatment of the disease in the last 2 months;
* Acute ischemic heart disease, unstable angina pectoris, exercise-induced ventricular arrhythmias, decompensated heart failure;
* History or suspicion of inability to cooperate properly in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Moderate to Vigorous Physical Activity (MVPA) | Baseline and after one-year of follow-up
  Total time in minutes spent in moderate- to-vigorous physical activity (MVPA) as measured by accelerometer
Change in Peak oxygen consumption (VO2peak) | Baseline and after one-year of follow-up
  VO2peak measured through of cardiopulmonary exercise test (CPET). Adjusted by anthropometrics measures and compared with reference values.

SECONDARY OUTCOMES:
Change in steps/day | Baseline and after one-year of follow-up
  Steps will be measured using a accelerometer by seven days. We will consider the mean of the measured period.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Blanco, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic, Barcelona, Spain